CLINICAL TRIAL: NCT04248595
Title: Clinical Study of Azacitidine Combined With Homoharringtonie Based Regimens in Acute Myeloid Leukemia
Brief Title: Study of Azacitidine Combined With Homoharringtonie Based Regimens in AML
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ge Zheng (Other)
Responsible Party: Sponsor-Investigator, Ge Zheng, Director of Department of Hematology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDYYGZ201912
Record Dates: First submitted 2020-01-22; First posted 2020-01-30 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Homoharringtonie; Azacitidine; Demethylation
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Homoharringtonine; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azacitidine plus HAG (Experimental): Patients of de novo or relapsed AML(age≥60y or ineligibility to receive intensive chemotherapy) will receive AZA+HAG (homoharringtonie, cytarabine, G-CSF) regiment as induction therapy. After complete remission(CR), the AZA+HAG regimen was further given 4-6 cycles and followed by azacitidine maintenance or until the disease progresses.
  AZA -Azacitidine HAG -Homoharringtonie, Cytarabine, G-CSF
  Interventions: Drug: Homoharringtonine; Drug: Azacitidine
- Azacitidine plus HIA (Experimental): Patients of de novo or relapsed AML(age<60y or eligible for intensive chemotherapy) will receive AZA +HIA(homoharringtonie, Idarubicin, cytarabine) regiments as introduction therapy. After CR, post-remission therapy will follow with NCCN guidelines.
  AZA -Azacitidine HIA -Homoharringtonie, Cytarabine, Idarubicin
  Interventions: Drug: Homoharringtonine; Drug: Azacitidine
- Azacitidine plus HDA (Experimental): Patients of de novo or relapsed AML(age<60y or eligible for intensive chemotherapy) will receive AZA +HDA(homoharringtonie, daunorubicin, cytarabine) regiments as introduction therapy., After CR, post-remission therapy will follow with NCCN guidelines.
  AZA -Azacitidine HDA -Homoharringtonie, Cytarabine, Daunorubicin
  Interventions: Drug: Homoharringtonine; Drug: Azacitidine

INTERVENTIONS:
Drug: Homoharringtonine — De novo AML or relapsed AML patients recieve chemotherapy regimen contained homoharringtonie and azacitidine.
  Other Names: HHT, Omacetaxine mepesuccinate
Drug: Azacitidine — De novo AML or relapsed AML patients recieve chemotherapy regimen contained homoharringtonie and azacitidine.
  Other Names: AZA

SUMMARY:
Rencent years have witnessed great progress of the treatment of acute myeloid leukemia (AML). However, most patients have poor outcomes following the currently first-line DA(daunorubicin, cytarabine)/IA(Idarubicin, cytarabine) chemotherapy, espiecially for the older patients and those not eligiable for receiving allo-HSCT. Azacitidine (AZA)，a hypomethylating agent, targets epigenetic gene silencing by inhibiting gene expression against malignant phenotypes and is currently approved to treat AML based on the NCCN guidelines. The homoharringtonie (HHT) could induce AML cell lines and primary myeloid leukemia cell apoptosis, and the effect was dose dependent. While, HHT could also induce leukemia cells to differentiate into normal state, eventually achieve the goal of treatment, and control the disease. The investigators conducted a clinical study to evaluate the efficacy and safety of the AZA plus HAG(homoharringtonie, cytarabine, G-CSF), HIA(homoharringtonie, Idarubicin, cytarabine)/HDA(homoharringtonie, daunorubicin, cytarabine). This study is aimed to demonstrate the efficacy and safety advantages of the regimens that cotain homoharringtonie and azacitidine.

DETAILED DESCRIPTION:
Currently, the treatment of acute myeloid leukemia (AML) still remains a therapeutic challenge. Patients received traditional chemotherapy have a low remission rate, poor prognosis and short survival for patients. New treatment strategies are needed in find out a better chemotherapy regimen.

Azacitidine (AZA), a hypomethylating agent, targets epigenetic gene silencing by inhibiting gene expression against malignant phenotypes. Azacitidine is currently approved to treat AML based on the NCCN guidelines. Novel combinations based on the azacitidine are currently undergoing, and the preliminary results brought promising hope to the treatment of AML.

The homoharringtonie (HHT) is a plant cytotoxic alkaloid derived from the trees of the genus Cephalotaxus. As a protein synthesis inhibitor, homoharringtonie plays a major role in the G1 / G2 phase in cells. In addition, it could induce AML cell lines and primary myeloid leukemia cell apoptosis, and the effect was dose dependent. Meanwhile it could also induce leukemia cells to differentiate into normal state, eventually controlled the progression of the disease.

Combination with azacitidine may become a new option.This study intends to apply azacitidine in combination with homoharringtonie for treating AML patients, aiming to improve the efficacy, reduce adverse events and improve the living qualities of patients.

Patients of de novo or relapsed AML(age≥60y or ineligibility to receive intensive chemotherapy) will receive AZA+HAG (homoharringtonie, cytarabine, G-CSF) regiment as induction therapy. After complete remission(CR), the AZA+HAG regimen was further given 4-6 cycles and followed by azacitidine maintenance or until the disease progresses.

Patients of de novo or relapsed AML(age<60y or eligible for intensive chemotherapy) will receive AZA +HIA(homoharringtonie, Idarubicin, cytarabine) or AZA+HDA(homoharringtonie, daunorubicin, cytarabine) regiments as introduction therapy. After CR, post-remission therapy will follow with NCCN guidelines.

The investigators choose historical AML patients receiving tranditional chemotherapy as a control group, to evaluate the efficacy and safety profiles.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnoised with acute myeloid leukemia
2. Meet the criteria of the 2016 WHO classification system(APL were excluded), based on blood cell counting, bone marrow biopsy, and cytogeneic diagnosis
3. Volunteered to sign the informed consent.

Exclusion Criteria:

1. Mental disorders or other conditions that cannot meet the requirements of research, treatment and monitoring
2. Uncontrolled cardiovascular disease
3. Allergic to azacytarine, homoharringtonie, or other drugs of this study
4. Any other conditions considered by the study investgators that are not suitable for participating in this clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
CR | From date of randomization or initial treatment until the date of first documented disease relapse from any cause，assessed up to 100 weeks.
  CR in months, in present of complete remission rate of all participants.

SECONDARY OUTCOMES:
Adverse events rates | From date of randomization or initial treatment until the end date of the study, assessed up to 100 weeks.
  Adverse events rates in percetage.
RFS | From date of randomization or complete remission until the date of first documented disease relapse from any cause，assessed up to 100weeks.
  RFS in months, in present of relapse free survival period of all participants
OS | From date of randomization until the date of first documented death from any cause or end of this study, whichever come first，assessed up to 100weeks.
  OS in months, in present of overall survival period of all participants

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Ge, M.D, Ph.D, Study Director — Medical School of South East University, China
Locations (1):
- Department of Hematology, Zhongda Hospital, Medical School of Southeast University, Nanjing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li J, Huang Y, Hou Y, Gu Y, Song C, Ge Z. High efficacy of azacitidine combined with homoharringtonine, idarubicin, and cytarabine in newly diagnosed patients with AML: A single arm, phase 2 trial. Front Oncol. 2022 Dec 8;12:1069246. doi: 10.3389/fonc.2022.1069246. eCollection 2022. PMID 36568250